CLINICAL TRIAL: NCT02874547
Title: Community Health Workers Using Patient Stories to Support Hypertension
Brief Title: Community Health Workers Using Patient Stories to Support Hypertension Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Warren Ferguson, Professor and Vice Chair, Department of Family Medicine and Community Health, University of Massachusetts, Worcester
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 5P60MD006912-02 (NIH)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Patients will receive five visits with a CHW during a 6 month period (two in-person and three by telephone). At the first visit, patients will meet the CHW who is trained in motivational interviewing techniques to deliver coaching to work on behavioral changes and introduce a 60 minute Digital Video Disc of five patient stories of individuals who have managed to control their hypertension.
  Interventions: Behavioral: Intervention
- Delayed Intervention (Other): Patients will receive print materials at time of consent and randomization. Four to six months after randomization, DI patients will receive an invitation to schedule an in-person visit at the health center to begin receiving the intervention protocol.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — During an in-person visit, patients receive a pamphlet in english and spanish and a storytelling Digital Versatile Disc (DVD) (developed for this project from interviews with hypertensive patients), supplemented by motivational interviewing delivered by the CHW. The CHW explores the patient's motivation to change associated with hypertension and counsels on risk factor control (tobacco, diet, physical activity). Patients receive a followup telephone call from the CHW in 2 weeks, 4 weeks, 2 months to support any changes or goals discussed at first visit. Six months after first intervention visit, patients are invited to schedule an in-person visit with the CHW at the health center to discuss goals and provide support for change.

SUMMARY:
Community Health Workers (CHWs) using patient stories to support hypertension management is a randomized controlled trial to evaluate the implementation of a CHW-delivered culturally appropriate storytelling intervention for english and spanish-speaking patients diagnosed with hypertension who receive care at community health center settings.

DETAILED DESCRIPTION:
Community Health Workers (CHWs) using patient stories to support hypertension (HTN) management is a CHW-delivered culturally appropriate storytelling intervention for patients diagnosed with HTN. We will develop and test interactive videos presenting stories of patients who have successfully made changes enhancing blood pressure control; and integrate this new tool with a CHW approach to management of hypertension. This two site, two-armed randomized controlled trial aims to recruit 252 english and spanish speaking patients with uncontrolled HTN. All participants are randomized to receive five visits (two in-person and 3 telephone calls) with CHWs either immediately (intervention condition (I)) or 6 months after enrollment (delayed intervention (DI)). Intervention participants receive the intervention immediately and DI participants receive print materials at enrollment and are telephoned 4-6 months after enrollment to schedule an in-person visit at the health enter to begin receiving the intervention protocol.

ELIGIBILITY:
Inclusion Criteria:

* English and Spanish speaking patients
* Male or female between the ages of 30 and 80
* Diagnosis of HTN and uncontrolled HTN, defined as (a) having an average systolic BP greater than or equal to 140 and /or diastolic BP greater than or equal to 90 over the past 12 months or (b) most recent BP reading within the previous 6 months as systolic BP greater than or equal to 140 and /or diastolic BP greater than or equal to 90.
* Willingness to be randomized to either intervention or delayed intervention

Exclusion Criteria:

* Pregnant women
* Patients planning to leave the Community Health Center in the next year
* Adults unable to consent

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2014-04-14 (Actual); Primary Completion 2016-09-14 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
changes in systolic and diastolic BP (SBP and DBP) | 6 months
  Entering SBP and DBP will be the most recent BP values in the 6 months before entry; exit BP values will be the average of two BP values taken at study exit.

SECONDARY OUTCOMES:
Reduce sodium intake | 6 months
  Self report of behavior change
Increased physical activity | 6 months
  Self report of behavior change
Greater medication adherence | 6 months
  Self report of behavior change
Blood Pressure maintenance | 12 months
  SBP and DBP will be the value obtained from the Electronic Health Record visit date 12 months after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Warren Ferguson, M.D., Principal Investigator — University of Massachusetts, Worcester
Locations (2):
- United States (2):
  - Lowell Community Health Center, Lowell, Massachusetts
  - Family Health Center of Worcester, Worcester, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Egan BM, Zhao Y, Axon RN. US trends in prevalence, awareness, treatment, and control of hypertension, 1988-2008. JAMA. 2010 May 26;303(20):2043-50. doi: 10.1001/jama.2010.650. PMID 20501926
- [Background] Ostchega Y, Dillon CF, Hughes JP, Carroll M, Yoon S. Trends in hypertension prevalence, awareness, treatment, and control in older U.S. adults: data from the National Health and Nutrition Examination Survey 1988 to 2004. J Am Geriatr Soc. 2007 Jul;55(7):1056-65. doi: 10.1111/j.1532-5415.2007.01215.x. PMID 17608879
- [Background] McWilliams JM, Meara E, Zaslavsky AM, Ayanian JZ. Differences in control of cardiovascular disease and diabetes by race, ethnicity, and education: U.S. trends from 1999 to 2006 and effects of medicare coverage. Ann Intern Med. 2009 Apr 21;150(8):505-15. doi: 10.7326/0003-4819-150-8-200904210-00005. PMID 19380852
- [Background] Swider SM. Outcome effectiveness of community health workers: an integrative literature review. Public Health Nurs. 2002 Jan-Feb;19(1):11-20. doi: 10.1046/j.1525-1446.2002.19003.x. PMID 11841678
- [Background] Houston TK, Allison JJ, Sussman M, Horn W, Holt CL, Trobaugh J, Salas M, Pisu M, Cuffee YL, Larkin D, Person SD, Barton B, Kiefe CI, Hullett S. Culturally appropriate storytelling to improve blood pressure: a randomized trial. Ann Intern Med. 2011 Jan 18;154(2):77-84. doi: 10.7326/0003-4819-154-2-201101180-00004. PMID 21242364
- [Derived] Hargraves JL, Bonollo D, Person SD, Ferguson WJ. A randomized controlled trial of community health workers using patient stories to support hypertension management: Study protocol. Contemp Clin Trials. 2018 Jun;69:76-82. doi: 10.1016/j.cct.2018.04.004. Epub 2018 Apr 12. PMID 29654929